CLINICAL TRIAL: NCT03011580
Title: Vitamin D3 to Enhance Resolution of Residual Pulmonary Inflammation in Patients Completing Antituberculosis Treatment (ResolveD-TB): a Proof-of-concept Intervention Study
Brief Title: Vitamin D to Resolve Inflammation After Tuberculosis (ResolveD-TB)
Acronym: ResolveD-TB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 011410
Record Dates: First submitted 2016-11-15; First posted 2017-01-05 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Tuberculosis
Keywords: Vitamin D
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate supplementation arm (Experimental): Fultium-D3 (oral cholecalciferol or vitamin D3) will be given at a dose of 9,600 IU/day for 8 weeks (three capsules once daily as each Fulitium D-3 capsules contains 3,200 IU vitamin D3). Participants may also be given a Sensemedic dispenser each for real-time adherence monitoring and shown how to use it.
  All participants will be given a supply of Fultium-D3 at a dose of 3,200 IU/day at the end of the study.
  Interventions: Dietary Supplement: Fultium-D3
- Delayed supplementation arm (Placebo Comparator): Oral placebo will be given for 8 weeks at a dose of three capsules once daily. Fultium-D3 and placebo will be identical in appearance and taste. Participants may also be given a Sensemedic dispenser each for real-time adherence monitoring and shown how to use it. All participants will be given a supply of Fultium-D3 at a dose of 3,200 IU/day at the end of the study.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fultium-D3 — Fultium-D3 (oral cholecalciferol or vitamin D3) will be given to participants in the immediate supplementation arm at a dose of 9,600 IU/day for 8 weeks at V2. At V3, all participants will be given a supply of Fultium-D3 at a dose of 3,200 IU/day.
  Arms: Immediate supplementation arm
Dietary Supplement: Placebo — 3 capsules of placebo will be given daily to participants in the delayed supplementation arm for 8 weeks at V2.
  Arms: Delayed supplementation arm

SUMMARY:
This Strategic Research Project is a translational proof-of-concept study that will determine whether vitamin D3 has potential to prevent recurrent tuberculosis (TB), as indicated by enhanced resolution of pulmonary inflammation detected using 18F-FDG PET-CT scanning. The extent of pulmonary inflammation detectable on PET-CT scanning is a validated biomarker that has previously been shown to predict risk of TB recurrence in patients taking anti-TB treatment. The investigators propose to explore whether vitamin D3 can enhance resolution of PET-CT-detectable pulmonary inflammation, on the basis of extensive preliminary data from in vitro studies and a Phase 2b clinical trial that the investigators have conducted, showing that high-dose vitamin D3 accelerates resolution of peripheral blood inflammatory responses in patients with pulmonary TB.

Forty vitamin D-deficient patients who have completed 6 months' TB treatment, but who still have residual pulmonary inflammation detectable on PET-CT scanning, will be allocated to receive either an 8-week course of high-dose oral vitamin D3 supplementation or placebo during the study period. The extent of pulmonary inflammation on PET-CT scanning will be compared between intervention vs. control groups at 8-week follow-up.

If the study shows a positive result, it will generate valuable proof-of-concept data that could be used to support an application to conduct a large phase 3 trial of vitamin D supplementation to prevent TB recurrence.

DETAILED DESCRIPTION:
Study design and its justification:

This is an exploratory study to compare the effects of vitamin D supplementation against placebo (capsules with no active drug) on residual pulmonary inflammation detectable with PET-CT scanning. If the study demonstrates that vitamin D supplementation can dampen down lung inflammation in patients who still have such inflammation at the end of antibiotic treatment, it will provide the basis for bigger and more rigorous studies. Half of the participants will be asked to take capsules containing vitamin D (the immediate supplementation group) and the other half placebo (the delayed supplementation group) for a duration of 8 weeks, once they have completed anti-tuberculosis treatment. There is an equal chance (1 in 2) that participants will be given either study medication - this allows the two groups to be fairly similar in background characteristics so that any differences in inflammation after 8 weeks would be put down to vitamin D supplementation.

The study will adopt a 'double-blind' approach, meaning that neither participants nor researchers will know which study medication each participant is taking for the duration of the study. This allows to minimise the influence that knowing the type of study medication each participant is taking might have on researchers' or participants' behaviour during the study, as these behaviours might affect the results of the study. This is also one of the reasons that the investigators have chosen to use placebo in this study, rather than comparing participants taking vitamin D to those who are not taking any study medication. In addition, the use of placebo may encourage participants to take the study medication. It is unlikely that the delay in starting vitamin D replacement for participants in the delayed supplementation arm would be harmful, as vitamin D deficiency is very unlikely to be associated with any acute medical problem, and the delay in its correction (8 weeks) is very short in relation to the likely duration of deficiency preceding the study, which is likely to have been longstanding (e.g. over years).

Study procedures:

* Attend up to three visits to hospital after they have completed a course of antibiotics for pulmonary tuberculosis. Visit 2 may be conducted via telephone with posting of study medication (by registered mail or courier)
* Take three capsules of study medication (each is 3,200 IU so a total of 9,600 IU) every day, using the dispenser provided by the investigators
* Give two blood samples: first =19 ml (~4 tsp), second =25 ml (~5 tsp)
* Give two coughing samples
* Have two chest PET-CT scans
* Receive five telephone calls, each lasting about five minutes
* Receive additional telephone calls if any doses are missed

Potential participants will be given a copy of the Patient Information Sheet (PIS) by a member of their usual care team at their scheduled clinic appointment after completing TB treatment and ample time (at least 24 hours) to decide whether they want to take part in the study. Those taking a PIS will be asked to complete a contact slip providing their contact details and authorising the research team to make contact with them once they have had a chance to read the information; this contact slip will be forwarded to the research team by the participant's usual care team.

Telephone call 1 - This will feed back results of tests of vitamin D status, calcium and renal function performed as part of usual care.

Potential participants who are found to be vitamin D deficient (serum 25[OH]D <50 nmol/L), normocalcaemic (serum corrected calcium <2.65 mmol/L) and to have eGFR >30 ml/min/1.73 m2 will be invited to attend Visit 1 (-2 weeks) for screening.

Visit 1 - Potential participants attending Visit 1 will be asked to give written informed consent to participate in the study. A PET-CT scan will be performed at the Department of Nuclear Medicine, Barts Health NHS Trust (radiation exposure for a PET-CT scan is 4.6 mSv). All women of childbearing age will be asked to do a urine pregnancy test before the PET-CT scan ; the scan will not proceed unless a negative pregnancy test result is obtained at this time. Blood samples (volume of 19 ml) for immunological testing and an induced sputum sample will also be taken during this visit. Participants' GPs will be notified by post about their involvement in the study at this stage, where consent has been given to do so.

Telephone call 2 - This will feed back results of tests of the PET-CT scan performed at Visit 1. Participants who are found to have significant residual PET-hot pulmonary inflammation on this scan (SUVmax ≥3 g/ml) will be invited to attend Visit 2 (0 weeks).

Visit 2 (0 weeks) - At this visit, eligible participants will be allocated to oral vitamin D replacement therapy at a daily dose of 9,600 IU of Fultium-D3 (cholecalciferol or vitamin D3) for 8 weeks for the immediate supplementation arm (n=20) or oral placebo for 8 weeks for the delayed supplementation arm (n=20). Fultium-D3 and placebo will be identical in appearance and taste and both will be given at a dose of three capsules once daily (each Fultium-D3 capsules contains 3,200 IU vitamin D3). Participants may also be given a CE-marked Sensemedic dispenser each for real-time adherence monitoring and shown how to use it. Participants will be advised of the symptoms of high blood calcium levels (nausea, vomiting, thirst, passing excessive amounts of urine or feeling generally unwell) and asked to contact a designated member of the study team if they develop these symptoms so that a blood test to check for high blood calcium levels can be arranged urgently. Any new symptoms reported between Visit 2 and Visit 3 will be assessed by a study doctor for potential association with the study medication. Arrangements will be made during this visit for telephone follow-up sessions. Visit 2 may be conducted via telephone with posting of study medication (by registered mail or courier) at an investigator's discretion.

Follow-up telephone calls (T3-5 and for missed doses) - Follow-up telephone calls will be made at 1 week (T3), 3 weeks (T4) and 5 weeks (T5) post-randomisation for all participants. A member of the study team will telephone participants at a pre-arranged time to check adherence to study medication and if there have been any problems with using the Sensemedic dispenser. Telephone calls will also be made to participants when a non-adherence is logged on the Sensemedic system. Additional intermediate study face-to-face visits will be arranged as necessary if any adherence issues are identified.

Visit 3 - PET-CT scans and measurement of whole blood (volume of 25 ml) and induced sputum inflammatory markers will be repeated at Visit 3 (+8 weeks). All women of childbearing age will be asked to do a urine pregnancy test before the PET-CT scan ; the scan will not proceed unless a negative pregnancy test result is obtained at this time. All radiological read-outs will be assessed by radiologists blinded to allocation, and compared between supplemented vs. unsupplemented patients using analysis of covariance to adjust for baseline values. All participants will be offered vitamin D supplementation after their 8-week follow-up assessment, prior to discharge from the study. Participants'GPs will be informed by post that their participation in the study has ended. All participants will be informed by post at the end of the study of whether they received vitamin D supplements or placebo between Visit 2 and Visit 3.

Discontinuation of study medication:

Participants whose study medication is discontinued will remain in follow-up as long as they consent to do so, and data will continue to be collected for them.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or more at enrolment
* Baseline serum 25-hydroxyvitamin D <50 nmol/L
* Maximum standardised uptake value (SUVmax) on baseline PET-CT ≥3 g/ml
* Completing antimicrobial therapy for pulmonary tuberculosis
* If a woman of child-bearing potential, has negative pregnancy test immediately prior to each PET-CT scan and agrees to use reliable form of contraception until she has completed the study
* Gives written informed consent to participate

Exclusion Criteria:

* Pregnant, breastfeeding or planning a pregnancy
* Baseline serum corrected calcium concentration ≥2.65 mmol/L
* Baseline eGFR ≤ 30 ml/min/1.73 m2
* Other contra-indication to vitamin D supplementation: known sarcoidosis, known hyperparathyroidism or known nephrolithiasis
* Taking concomitant phenytoin, barbiturate, cardiac glycoside, oral glucocorticoid or vitamin D supplement
* Known allergy to vitamin D or its excipients
* Currently taking part in another interventional research study
* PET-CT scan within the previous 6 months
* Any inclusion criteria not met

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Mean maximum standardised uptake value (SUVmax) on PET-CT scanning at 8-week follow-up. | 8 weeks in total

SECONDARY OUTCOMES:
Inflammation Score on PET-CT at 8-week follow-up. | 8 weeks in total
  A single composite outcome score derived from the following components: total glycolytic activity, total cavitary air, total volume of lesions with radiodensity ranging from -100 to +200 Houndsfield Units
Proportion of PET-hot lesions resolving over the course of the study | 8 weeks in total
Total and differential white cell counts | 8 weeks in total
Concentrations of inflammatory mediators in serum at 8-week follow-up. | 8 weeks in total
Concentrations of inflammatory mediators in plasma at 8-week follow-up. | 8 weeks in total
Concentrations of inflammatory mediators in induced sputum supernatants at 8-week follow-up. | 8 weeks in total
Concentrations of inflammatory mediators in supernatants of antigen-stimulated whole blood at 8-week follow-up. | 8 weeks in total
Induced sputum transcriptional profiles at 8-week follow-up. | 8 weeks in total
Whole blood transcriptional profiles at 8-week follow-up. | 8 weeks in total
Sputum microbiology at 8-week follow-up. | 8 weeks in total
  To assess the proportion of samples in which Mycobacterium tuberculosis can be detected after 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Martineau, Prof, Principal Investigator — Barts and The London School of Medicine and Dentistry, Queen Mary University, University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available. Non-patient identifiable data will be presented in paper, abstract and presentation to conferences.